CLINICAL TRIAL: NCT05679349
Title: Provider Support and Patient Outreach in Lung Cancer Screening
Brief Title: Support and Outreach to Increase Screening for Lung Cancer in Patients With a History of Smoking
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ronald Myers (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ronald Myers, Professor - Medical Oncology, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Screening
Other Study IDs: 22F.808; R01CA258849 (NIH); JT 24704 (Other: JeffTrial Number)
Record Dates: First submitted 2022-12-23; First posted 2023-01-11 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Lung Carcinoma; Tobacco-Related Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Providers): (survey, online educational activity) (Experimental): Participants complete survey on study. Participants undergo online educational activity on study. Participants undergo distance learning on study.
  Interventions: Other: Survey Administration; Other: Educational Activity
- Group B (Providers): (survey) (Active Comparator): Participants complete survey at baseline and end of study survey.
  Interventions: Other: Survey Administration
- Group A (Patients): (EHR, educational activity, counseling)) (Experimental): Patients undergo EHR review on study. Patients undergo educational activity on study. Patients also undergo SDM counseling once on study.
  Interventions: Other: Electronic Health Record Review; Other: Educational Activity; Other: Counseling
- Group B (Patients): (survey) (Active Comparator): Patients undergo EHR review on study and complete telephone survey throughout the trial.
  Interventions: Other: Survey Administration; Other: Electronic Health Record Review

INTERVENTIONS:
Other: Survey Administration — Complete survey
  Arms: Group A (Providers): (survey, online educational activity)
Other: Educational Activity — Undergo online shared decision making training and distance learning
  Arms: Group A (Providers): (survey, online educational activity)
Other: Survey Administration — Complete survey
  Arms: Group B (Providers): (survey)
Other: Electronic Health Record Review — Undergo electronic health record review
  Arms: Group A (Patients): (EHR, educational activity, counseling))
Other: Educational Activity — Undergo online shared decision making training and distance learning
  Arms: Group A (Patients): (EHR, educational activity, counseling))
Other: Counseling — Undergo shared decision making counseling
  Other Names: Counseling Intervention
  Arms: Group A (Patients): (EHR, educational activity, counseling))
Other: Survey Administration — Complete survey
  Arms: Group B (Patients): (survey)
Other: Electronic Health Record Review — Undergo electronic health record review
  Arms: Group B (Patients): (survey)

SUMMARY:
This clinical trial tests how well providing education improves screening for lung cancer in patients with a history of smoking. Screenings may help doctors find lung cancer sooner when it may be easier to treat. Education and counseling may be an effective method to help providers and patients learn about lung cancer screening. Providing education and decision counseling to providers and patients may increase lung cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess intervention impact on lung cancer screening (LCS). II. Assess intervention impact on shared decision making (SDM).

SECONDARY OBJECTIVES:

I. Identify mediators and moderators of LCS. II. Assess intervention implementation barriers and facilitators.

EXPLORATORY OBJECTIVES:

I. Assess intervention impact on:

Ia. LCS referral; Ib. Tobacco treatment services referral; Ic. Repeat annual LCS among participants with a normal initial screening result; Id. Follow-up diagnostic evaluation for participants with an abnormal screening result.

OUTLINE: Providers are randomized to 1 of 2 groups. Patients are randomized to 1 of 2 groups.

PROVIDERS:

GROUP A: PROVIDER SUPPORT GROUP: Participants complete survey on study. Participants undergo online educational activity on study. Participants undergo distance learning on study.

GROUP B: PROVIDER CONTROL GROUP: Participants complete survey at baseline and end of study survey.

PATIENTS:

GROUP A: Patients undergo electronic health records (EHR) review on study. Patients undergo educational activity on study. Patients also undergo SDM counseling once on study.

GROUP B: Patients undergo EHR review on study and complete telephone survey throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* PRACTICE LEVEL:
* Primary care practice (family medicine, geriatrics, internal medicine) in one of the 4 participating health systems
* Practice using the main electronic medical record (EMR) of each system, in order to run appropriate patient recruitment reports
* Practice with at least 50% of practice providers (physicians and advanced care providers) consenting to participate
* PATIENT LEVEL:
* Have an office or telemedicine established patient visit scheduled with a primary care provider in one of the participating practices within next 14 to 25 days
* 50 to 77 years of age
* Have at least a 20-pack-year smoking history (based on self-report at baseline eligibility assessment)
* Currently smoke or have quit smoking within the past 15 years (based on self-report at baseline eligibility assessment)
* Able to communicate in English or Spanish (determined at baseline eligibility assessment)

Exclusion Criteria:

* PATIENT OUTREACH:
* Any lung computed tomography (CT) or low-dose computed tomography (LDCT) scan in the past 11 months, current procedural terminology (CPT) Codes are as follows

  * G0297 - LDCT screening
  * 71250 - CT w/o contrast
  * 71260 - CT w/ contrast
  * 71270 - CT with and w/o contrast
  * 71275 - CT angiography chest
  * 78815 - Positron emission tomography computed tomography (PET CT) skull base to mid-thigh
  * 78816 - PET CT whole body
* Prior history of lung cancer (The patient's problem list includes a problem with an international classification of diseases (ICD10) code of "Z85.118" or one beginning with "C34.", or by self-report at baseline eligibility assessment)
* Recent hospitalization (Admission date within the last 60 days listed in electronic health record (EHR), or by self-report at baseline eligibility assessment)
* Dementia (diagnosis codes F03.90 or F03.91) in EHR

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 822 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Completion of initial lung cancer screening (LCS) | Within 4 months of randomization
  LCS will be assessed through an endpoint electronic medical records (EMR) search, supplemented with a question on the participant endpoint survey to capture any LCS performed outside the health system and/or not captured in the EMR.

SECONDARY OUTCOMES:
Referral for LCS | Up to 5 years
  Referrals for lung cancer screenings will be found by reviewing electronic medical records.
Tobacco cessation services | Up to 5 years
  Referrals for tobacco treatment services will be found by reviewing medical records.
Repeat annual lung cancer screenings within 11-16 months of original screening | within 11-16 months of original screening
  Number of repeat screenings will be found by reviewing electronic medical records.
Diagnostic follow up after initial lung cancer screening | Up to 4 months of screening
  Number of patients that had follow up within 4 months of initial lung cancer screening will be found by reviewing electronic medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States